CLINICAL TRIAL: NCT00724139
Title: The Effect of Training With Custom-Made Biomechanical Perturbation Platform on Kinetics, Kinematics and Electromyography in Knee Osteoarthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: protocol # 078
Record Dates: First submitted 2008-07-27; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- 1 (Experimental): patients (aged 50-75) with Symptomatic knee OA for at least 6 months, fulfilled American College of Rheumatology clinical criteria for OA of the knee and radiographically assessed osteoarthritis of the knee graded 1-2 according to the Kellgren & Lawrence scale.
  Interventions: Device: : APOS biomechanical gait system, Apos - Sports and Medical Technologies Ltd. Hertzlia, Israel

INTERVENTIONS:
Device: : APOS biomechanical gait system, Apos - Sports and Medical Technologies Ltd. Hertzlia, Israel — training program utilizing a novel biomechanical system comprising four modular elements attached onto foot-worn platforms which conveys perturbation throughout the gait cycle

SUMMARY:
The aim of this study is to evaluate the outcome of specific repetitive biomechanical perturbation training on motor patterns.

The first hypothesis of this project is that footwear derived biomechanical challenges will convey active and passive matching biomechanical responses (i.e. kinetic, kinematic and electromyographic) trough out the musculoskeletal kinematic chain.

The second hypothesis of the project is that repetitive exposure to in-situ (trough out the gait sickle) introduction to a biomechanical stimulus would generate a process of motor learning thus conveying plasticity of existing locomotor patterns and gait strategies.

DETAILED DESCRIPTION:
Design: Prospective, case control Setting: subjects will undergo a tailored training program utilizing a novel biomechanical system comprising four modular elements attached onto foot-worn platforms (APOS system, Apos - Sports and Medical Technologies Ltd. Hertzlia, Israel) which conveys perturbation throughout the gait sickle. Pre and post training level walking will be examined via: (1) a three-dimensional motion analysis system and (2) ground reaction force analysis using force platforms (3) Electro-Myography system. Each subject will be examined in 4 different settings Patients will then participate in continued biomechanical perturbation training for 3-6 month and will then undergo a second gait examination Ages Eligible for Study: 50 Years - 75 Years, Genders Eligible for Study: None Accepts patients suffering from medial compartment knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Community-dwelling older adults.
  2. Symptomatic knee OA for at least 6 months, fulfilled American College of Rheumatology clinical criteria for OA of the knee and radiographically assessed osteoarthritis of the knee graded 1-2 according to the Kellgren & Lawrence scale.
  3. Ambulatory and active patients that can precipitate the gait analysis.
  4. Age 50-75.
  5. No prior joint replacement in the lower extremity.

Exclusion Criteria:

* Exclusion Criteria:

  * Knee pain due to pathologic conditions other than OA, such as rheumatoid arthritis and pseudogout.
  * Knee with flexion contracture greater than 20°.
  * Patients with hip problems, symptomatic lumbar spine disease, spinal cord.
  * Ataxic gait related to neurologic disease.
  * Patients with increased tendency to fall.
  * Lack of physical or mental ability to perform or comply with the treatment procedure.
  * Diabetes mellitus.
  * History of pathological osteoporotic fracture.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
footwear derived biomechanical challenges will convey active and passive matching biomechanical responses (i.e. kinetic, kinematic and electromyographic) trough out the musculoskeletal kinematic chain | 6 months

SECONDARY OUTCOMES:
would repetitive exposure to in-situ (trough out the gait sickle) introduction to a biomechanical stimulus would generate a process of motor learning | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Technion Israel institute of technology, Haifa, Israel

REFERENCES:
- [Derived] Debbi EM, Wolf A, Goryachev Y, Rozen N, Haim A. Alterations in sagittal plane knee kinetics in knee osteoarthritis using a biomechanical therapy device. Ann Biomed Eng. 2015 May;43(5):1089-97. doi: 10.1007/s10439-014-1177-3. Epub 2014 Nov 7. PMID 25377767